CLINICAL TRIAL: NCT03046082
Title: Anaerobic Antibiotic Usage for Pneumonia in the Medical Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Jeffrey Jennings, Staff Physician, Henry Ford Health System
Other Study IDs: 10229
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antibiotics — Observation of antibiotic types given to patients with pneumonia.

SUMMARY:
Observation of prescription usage of anaerobic antibiotics for patients admitted to the ICU with pneumonia.

DETAILED DESCRIPTION:
Pneumonia is a common admitting diagnosis in the intensive care unit (ICU). When aspiration is suspected, antibiotics to cover anaerobes are frequently used , but in the absence of clear risk factors, current guidelines have questioned their role. It is unknown how frequently these guidelines are followed.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients with diagnosis of pneumonia

Exclusion Criteria:

* patients with abdominal infections such as c diff.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the intensive care unit with a diagnosis of pneumonia.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Usage of anaerobic antibiotics | 6 months
  Percent of patients receiving inappropriate anaerobic antibiotics

IPD SHARING:
Plan to Share IPD: Undecided